CLINICAL TRIAL: NCT02270762
Title: Effect of Early Passive Verticalization in Pulmonary Recruitment Evaluated With Electric Impedance Tomography
Brief Title: Early Passive Verticalization in Critically Ill Patients
Acronym: TILT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Early passive verticalization
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Critical Illness
Keywords: Early Physical Exercise; Early Passive Exercise; Alveolar Recruitment; Electrical Impedance Tomography; Oxygenation; Ventilation
MeSH Terms: conditions — Critical Illness; Motor Activity; Respiratory Aspiration | interventions — RE1-silencing transcription factor; Beds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1) Rest in bed (Experimental): First evaluation of EIT with patient in bed at 30º of head inclination during 5 minutes.
  Interventions: Other: Rest in bed
- 2) Passive Verticalization (Experimental): Second evaluation of EIT with patient in tilt table at 60º of verticalization during 10 minutes.
  Interventions: Other: Passive verticalization
- 3) Rest in bed (Experimental): Last evaluation of EIT with patient in bed at 30º of head inclination during 20 minutes.
  Interventions: Other: Rest in bed

INTERVENTIONS:
Other: Rest in bed
  Other Names: Basal position
  Arms: 1) Rest in bed
Other: Passive verticalization
  Other Names: Tilt Table; Early Passive verticalization; Early Assisted verticalization; Early physical therapy; Early physiotherapy
  Arms: 2) Passive Verticalization
Other: Rest in bed
  Other Names: Basal position
  Arms: 3) Rest in bed

SUMMARY:
In the critically patient bed rest and inmovilization are some of the responsable of the development of respiratory complications. Early physical exercise is a tool to prevent respiratory complications as lost of respiratory muscle strength, decrease in functional residual capacity and hypoxemia improving oxygenation. In some cases critically ill conditions implies use of pharmacological sedation. That condition limit the active physical exercise. However, some technicals aids as Tilt table allows execution of passive early movilization.

The aim of this study is to assess the effect of early passive verticalization assisted by tilt table on alveolar recruitment and pulmonary ventilation in intensive care unit (ICU) patients, evaluated with electrical impedance tomography (EIT) ICU patients included at day of evaluation will be evaluated consecutively with EIT in three stages; 1) in the supine position (at 30° of inclination), 2) verticalized in tilt table (at 60º of inclination) 3) in the supine position (at 30° of inclination)

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted at the Intensive Care Medical/Sirurgical Unite of Clinic Saint Luc
* Days of hospitalization between 1 and 10
* Hemodynamically stable
* Patient or family member sign the informed consent
* Sedated patients

Exclusion Criteria:

* With risk of evisceration
* Therapy withdrawal
* With cardiac devices (Pace Maker)
* Persistent cough
* Patches or open wounds in zone of electrodes
* Presence of high vasopressor medication (noradrenaline > 3 mg/h)
* PEEP > 15 cm H2
* Acute Myocardial Infarction
* Active bleeding
* Intracranial pressure > 20 mm Hg or with major inestability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary electric impedance tomography (EIT) before, during and after single session of early passive verticalization | Meassure of EIT during 10 minutes of early passive verticalization and will compared with baseline EIT
  The change in pulmonary recruitment will be evaluated with electrical impedance tomography (EIT) in single session of early passive verticalization. First measure will be made for five minutes with EIT, in bed; second measure will be made during passive verticalization for ten minutes with EIT and last measure will be made after verticalization for twenty minutes with EIT. All impedanciometries obtained in the patient in different activities will compare each.
Change in PaO2 before, during and after single session of early passive verticalization | Meassure of PaO2 after 20 minutes of passive verticalization and will compared with baseline PaO2
  Before passive verticalization will be taken a sample of arterial blood gases for determinate the initial PaO2 of the patient. Twenty minutes after passive verticalization will be taken a new sample of arterial blood gases to establish the diference between PaO2 before verticalization and after verticalization

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Meaux, PT, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Cheryl E Hickmann, PT, PhD student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Jean Roeseler, PT, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Pierre-François Laterre, MD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc)
Locations (1):
- Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc), Brussels, Belgium